CLINICAL TRIAL: NCT01450722
Title: Paclitaxel Eluting Stent in Long Superficial Femoral Artery Obstruction: a Prospective, Randomized Comparison With Bypass Surgery Using PTFE Graft in a Finnish Multicenter Study
Brief Title: Paclitaxel Eluting Stent in Long SFA Obstruction: A Prospective, Randomized Comparison With Bypass Surgery
Acronym: finnptx
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Tampere University Hospital (Other); Oulu University Hospital (Other); Finnish Society of Interventional radiology (Unknown); North Karelia Central Hospital (Other); Paijat-Hame Hospital District (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5063524
Record Dates: First submitted 2011-10-07; First posted 2011-10-12 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Chronic Lower Limb Ischemia; Peripheral Athero Obstructive Disease; Critical Ischemia; Claudication
Keywords: Chronic lower limb ischemia; claudication; chronic critical ischemia
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- drug eluting stent (Active Comparator): Paclitaxel eluting stent for long superficial femoral artery obstruction
  Interventions: Procedure: bypass surgery, stent placement; Procedure: stent placement
- bypass operation (Active Comparator): femoropopliteal artery bypass operation by using synthetic PTFE graft
  Interventions: Procedure: bypass surgery, stent placement

INTERVENTIONS:
Procedure: bypass surgery, stent placement — bypass surgery, stent placement
  Other Names: PTX stent
Procedure: stent placement — placement of paclitaxel eluting stent in long superficial femoral artery obstruction
  Other Names: PTX Cook
  Arms: drug eluting stent

SUMMARY:
Chronic lower limb ischemia due to atherosclerosis causes significant morbidity especially in elderly: the prevalence of asymptomatic obstructive peripheral atherosclerosis among 40-74 old is 4-22%. The prevalence of its milder symptomatic manifestation, intermittent claudication among 40 years old men is about 1% and among 70 years old it is 7%. In about 10% of the patients the ischemia worsens to threat the vitality of the limb. Although intermittent claudication has a benign prognosis and can often treated conservatively, more severe forms with extensive arterial obstructions require revascularization, either open surgical or endovascular. Surgical bypass operations are currently the standard reference for treating long femoral artery obstructions. Surgical bypass operations are accompanied by significant acute complications and late adverse effects, especially in patients with associated cardio-cerebrovascular and pulmonary diseases, and less invasive, safe, and effective endovascular therapies are seeked for. The long term patency rates of infrainguinal balloon angioplasty (PTA) vary largely in different studies but they are mostly poor when long femoral arterial obstructions have been treated. Drug eluting stents have shown great promise in coronary artery interventions. The purpose of this study is to compare Paclitaxel eluting Zilver PTX nitinol stent (Cook INC) with bypass surgery using PTFE graft to proximal popliteal artery in the treatment of long femoral artery obstructions (total length of 10-25 cm) in a prospective, randomized, Finnish multi center trial with consecutive claudicant and chronic critical ischemia patients. The aim is to randomize altogether 400 patients during about two years in five universities and in 2-3 central hospitals. The primary end point is patency at 24 month follow up. Secondary end points are primary success at patient discharge, complications, 30-day mortality, target lesion revascularization, quality of life, and economical analysis.

DETAILED DESCRIPTION:
BACKGROUND Chronic lower limb ischemia due to atherosclerosis causes significant morbidity especially in elderly: the prevalence of asymptomatic obstructive peripheral atherosclerosis among 40-74 old is 4-22%. The prevalence of its milder symptomatic manifestation, intermittent claudication among 40 years old men is about 1% and among 70 years old it is 7%. In about 10% of the patients the ischemia worsens to threat the vitality of the limb. Although intermittent claudication has a benign prognosis and can often treated conservatively, more severe forms with extensive arterial obstructions require revascularization, either open surgical or endovascular. Surgical bypass operation is currently the standard reference for treating long SFA obstructions. Up to 81% two-year patency can be appreciated after bypass with a good quality sapheneous vein. If synthetic graft is used the long term patency is somewhat lower, up to 67% according to a systematic review (Klinkert et al 2004).

The long term patency rates of infrainguinal balloon angioplasty (PTA) vary largely in different studies. At 1 year, primary patency rates of 47% to 86%, at three years 27% to 69%, and at six years 23% to 36% are reported in the literature. Highly variable and mostly poor patency rates, between 22 to 64% at 6-12 months have been reported by using subintimal angioplasty for the treatment of femoral and femoropopliteal lesions. (Met et al. 2008) In the femoropopliteal region, highly variable 1-year primary patency rates between 22% and 81% with various stents have been reported (Matsi et al 1994, Sapoval et al 1992, Grimm et al 2001, Lugmayr et al 2002). In three randomised studies, although the primary success rate of stent placement was higher than that after balloon angioplasty alone, the long-term patency was not improved by using stents (Cejna et al 2001, Grimm 2001). A meta-analysis revealed similar patency rates after balloon dilation and stent implantation (34). The authors of the largest randomized multicenter comparison of femoropopliteal PTA and balloon expanded stent placement with 154 treated limbs summarised that the beneficial effect of stents is to rescue PTA failures (54). In one study three year primary patency rate of 76% was obtained after primary stenting of relatively short, less than 6 cm long lesions (Lugmayr et al 2002). However, midterm restenosis after long-segment femoropopliteal stenting remains a problem. In recent single-center observational study in which long segments (median length 16 cm) were covered by nitinol stent after initial failure of PTA, the primary patency was only 54% at one year. Stent in the femoropopliteal artery are exposed to unique long term stress in the form of repeated compression, flexion and torsion and it is probably the reason why recent studies have revealed stent fractures in up to 50% of nitinol stents 1 year after placement (Schneinert et al 2005) and in 19% of Wallstents a mean of 43 months after placement (Sclager et al 2005). The fractures seem to be associated with poorer patency and they are more common in longer stents.

Drug eluting stents have shown great promise in coronary artery interventions. One of these drugs, sirolimus, that is a natural macrocyclic lactone with potent immunosuppressive and antimitotic action, has been tried also at femoral arteries. Sirolimus-eluting self-expanding nitinol SMART stent was compared in a small (57 patients) randomized, double-blind multi-center study with the bare metal stent (SIROCCO II trial) in treating femoral artery lesions with average length of 8 cm (Duda et al 2005). Exceptionally low angiographically verified binary restenosis rate of 7.7% was registered at the bare metal stent group. Although the restenosis rate was zero and there was less mean late loss in diameter in the drug stent group the difference did not reach statistical difference.

Paclitaxel is a mitotic inhibitor and another antiproliferative agent and widely used, effective agent in drug eluting stents to reduce restenosis in coronary circulation. Paclitaxel binds specifically to the beta-tubulin subunit of microtubules and appears to antagonize the disassembly of this key cytoskeletal protein; this action results in accumulation of microtubule bundles and aberrant microtubular derived structures in the mitotic phase of the cell cycle. Zilver PTX (Cook Medical) paclitaxel-eluting stent is designed for the SFA. It is a nitinol stent coated with paclitaxel only, with no polymer or binder. A recent prospective, randomized trial reported significantly better 24-month event-free survival among patient receiving PTX stent than among those treated with PTA (86,6% vs. 77.6%, p<0.01). Primary patency at 24 months of the PTX stent group was 74.8% vs 32.4% for the PTA group. (Dake , LINC 2011).

PURPOSE AND STUDY RATIONALE

To compare Paclitaxel eluting Zilver PTX stent (Cook INC) with bypass surgery using PTFE graft to proximal popliteal artery in the treatment of long SFA obstructions in a prospective, randomized, Finnish multi center trial with consecutive claudicant and chronic critical ischemia patients. Bypass with a synthetic graft instead of autogeneous vein is used as a reference standard because of the difficulty to standardize the quality of available vein and because the bypass done to the proximal popliteal artery with the graft types gives very similar results. The aim is to randomize altogether 400 patients during about two years in five university and in 2-3 central hospitals.

The power analysis of study is based on non-inferiority hypothesis, i.e. to show that paclitaxel eluting stent is not inferior to bypass surgery in 24 month patency. With accepted marginal for equality 5%, assuming surgical group patency 75% and non-inferiority margin 10% and using 1:1 randomization the sample size for a power of 80% to detect non-inferiority of the test treatment is 590 (295/295).

PATIENT RECRUITMENT

Consecutive patients fulfilling the inclusion criteria will be asked to the study by vascular surgeon or interventional radiologist after the diagnostic imaging study. A consensus of a vascular surgeon and interventional radiologist is required: for an elective patient this is acquired in a weekly vascular meeting and for an urgent patient by consultation. The patient will be provided no additional compensation for participation but normal travel expenses for clinical visits will be paid. The patient's identity and personal study data will be available only for the researchers of the trial. Normal clinical patient insurance is applied.

PREOPERATIVE IMAGING AND VASCULAR LAB

MR-angio, CT angio, or catheter angio (DSA) is performed for planning of the therapy.

Ankle brachial index is measured..

INTERVENTIONS

Balloon angioplasty is performed before and after stent placement. Stenting is done from healthy-to-healthy segment.

Surgery is performed by using PTFE graft with distal distal anastomosis at above knee popliteal artery.

POSTOPERATIVE MEDICATION

Stent group: ASA 100 mgx1, Simvastatin , Clopidogrel 300 mgx1, 75 mgx1 for 6 months

Surgery: ASA 100 mgx1, Simvastatin

POSTOPERATIVE FOLLOW- UP

AB-index and duplex ultrasound study will be performed at patient discharge. Clinical visit to a vascular surgeon is scheduled at 1, 6, 12, and 24 months with Ankle-brachial index measurement and duplex US study.

STUDY COORDINATION AND MONITORING

The main investigator of the trial is professor Hannu Manninen, Kuopio University Hospital. The other investigators in KUH are M.Ds. Kimmo Mäkinen, Petri Saari, and Jussi Kärkkäinen. The main investigator in Helsinki, Oulu, Tampere, and Turku University Hospitals are Jukka Perälä, Kimmo Lappalainen, Janne Korhonen, and Riitta Rautio, correspondingly. Randomization is performed centralized by a study coordinator (Marja-Liisa Sutinen, Kuopio) Analysis of imaging studies is performed in a core lab. The trial will possibly be monitored, which will be performed by an authorized person and coordinated by the research unit of Kuopio University Hospital.

STUDY ENDPOINTS

Study end points are determined according to CIRSE/SVS standards. Primary endpoint: Patency at 24 month follow-up by objective means with the aid of AB-index measurement and duplex US measurement.

Secondary endpoints:

Primary success and assisted primary success is registered at patient discharge.

Complications classified as minor and major. 30-day mortality. Target lesion revascularization (TLR), which was defined as any revascularization procedure, percutaneous or surgical, involving the target lesion.

AFS (amputation free survival) Economical analysis of direct and indirect costs. Life quality analysis.

DATA ANALYSIS

Randomization will be performed and coordinated by a common research coordinator for all participating centers. Imaging data will be archieved to a secured science PACS of Kuopio University Hospital and the image analysis will be performed by an independent researcher without knowledge of the patient data.

Primary procedural success and complications are defined according to established EVS/CIRSE guidelines. Cumulative patency rate will be calculated by Kaplan-Meier method and the statistical difference between the survival curves will be determined by the means of log-rank test. Quality of life analysis will be done using RAND-36 questionnaire.

BUDGET

Study coordinator will be recruited for 12 months. EVO funding will be applied.

TIME SCHEDULE

Approval of ethical committee in Kuopio: May 2011, in other centers August 2011.

Patient interventions start June 2011, cathering until December 2013. End of Follow up December 2015.

PUBLICATION PLAN

The sresults will be published in 2 - 3 original publications international peer reviewed journals and they will be a main portion of one Thesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from severe life-style limiting claudication indicating revascularization as well as patients suffering from chronic critical ischemia and having de-novo SFA obstruction with total length of 7-20 cm will be recruited.
* For claudicant patients an attempt of conservative treatment should be attempted before revacularization therapy. Both surgical bypass operation and endovascular treatment should be able to be safely performed;
* the patient has not extensive additional cardio-pulmonary and/or cerebro-vascular diseases increasing remarkably operative risk.
* At least one patent artery is to the ankle level.
* The patient has given his/her informed consent.
* Previous or simultaneus endovascular therapy of coexisting iliac disease is not a contraindication but study groups should be balanced.
* Unplanned common femoral artery endarterectomy is not a contraindication when it is done at the same intervention to facilitate anastomosis creation.

Exclusion Criteria:

* Patients who have not given their written informed consent.
* Patient has allergy for iodine contrast agent.
* Patient is undergoing hemodialysis.
* Patient has undergone previous endovascular treatment for the target lesion (restenotic lesions).
* Patient has also infrapopliteal disease indicating revascularization.
* Patient is pregnant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-10; Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary patency of the stent or graft at two year follow up | Ultrasound study at 2 years

SECONDARY OUTCOMES:
Amputation free survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hannu I Manninen, Professor, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

REFERENCES:
- [Derived] Bjorkman P, Auvinen T, Hakovirta H, Romsi P, Turtiainen J, Manninen H, Venermo M. Drug-Eluting Stent Shows Similar Patency Results as Prosthetic Bypass in Patients with Femoropopliteal Occlusion in a Randomized Trial. Ann Vasc Surg. 2018 Nov;53:165-170. doi: 10.1016/j.avsg.2018.04.014. Epub 2018 Jun 7. PMID 29886215